CLINICAL TRIAL: NCT01216761
Title: Blood Culture Contamination: A Cluster-randomized Cross-over Trial Evaluating the Comparative Effectiveness of Three Skin Antiseptic Interventions
Brief Title: A Cluster-randomized Cross-over Trial Evaluating the Comparative Effectiveness of Three Skin Antiseptic Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Laraine Washer, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: N010316 - 1932.II
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Bacteremia
Keywords: Bacteremia; Blood culture; Contamination; Antiseptic agents
MeSH Terms: conditions — Bacteremia | interventions — chlorhexidine gluconate; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHG then PI then IT (Active Comparator): Skin antisepsis prior to any peripheral blood culture collection on Floor A was performed with CHG for 3 months, followed by PI for 3 months, followed by IT for 3 months. Each 3 month intervention period was separated by a one month wash out period where data regarding blood culture contamination was not collected.
  2% chlorhexidine gluconate/70% isopropyl alcohol packaged in a single 1.5 ml Frepp applicators (Enturia, Leewood KS) -- CHG
  10% povidone iodine aqueous solution packaged in a single 0.67 Sepp applicator (Enturia, Leewood KS) -- PI
  Iodine tincture (2% iodine and 2% sodium iodide diluted in 50% ethanol) packaged in a single 0.67 mL Sepp applicator (Enturia, Leewood KS) -- IT
  Interventions: Drug: Iodine tincture; Drug: Chlorhexidine gluconate; Drug: Povidone iodine
- IT then CHG then PI (Active Comparator): Skin antisepsis prior to any peripheral blood culture collection on Floor B was performed with iodine tincture for 3 months, followed by Chlorhexidine gluconate for 3 months, followed by povidone iodine for 3 months. Each 3 month intervention period was separated by a one month wash out period where data regarding blood culture contamination was not collected.
  Iodine tincture (2% iodine and 2% sodium iodide diluted in 50% ethanol) packaged in a single 0.67 mL Sepp applicator (Enturia, Leewood KS) -- IT
  2% chlorhexidine gluconate/70% isopropyl alcohol packaged in a single 1.5 ml Frepp applicators (Enturia, Leewood KS) -- CHG
  10% povidone iodine aqueous solution packaged in a single 0.67 Sepp applicator (Enturia, Leewood KS) -- PI
  Interventions: Drug: Iodine tincture; Drug: Chlorhexidine gluconate; Drug: Povidone iodine
- PI then IT then CHG (Active Comparator): Skin antisepsis prior to any peripheral blood culture collection on Floor C was performed with povidone iodine for 3 months, followed by iodine tincture for 3 months, followed by chlorhexidine gluconate for 3 months. Each 3 3 month intervention period was separated by a one month wash out period where data regarding blood culture contamination was not collected.
  10% povidone iodine aqueous solution packaged in a single 0.67 Sepp applicator (Enturia, Leewood KS) -- PI
  Iodine tincture (2% iodine and 2% sodium iodide diluted in 50% ethanol) packaged in a single 0.67 mL Sepp applicator (Enturia, Leewood KS) -- IT
  2% chlorhexidine gluconate/70% isopropyl alcohol packaged in a single 1.5 ml Frepp applicators (Enturia, Leewood KS) -- CHG
  Interventions: Drug: Iodine tincture; Drug: Chlorhexidine gluconate; Drug: Povidone iodine

INTERVENTIONS:
Drug: Iodine tincture — Iodine tincture (2% iodine and 2% sodium iodide diluted in 50% ethanol) packaged in a single 0.67 mL Sepp applicator (Enturia, Leewood KS)
Drug: Chlorhexidine gluconate — 2% chlorhexidine gluconate/70% isopropyl alcohol packaged in a single 1.5 ml Frepp applicators (Enturia, Leewood KS)
Drug: Povidone iodine — 10% povidone iodine aqueous solution packaged in a single 0.67 Sepp applicator (Enturia, Leewood KS)

SUMMARY:
Background: Contaminated blood cultures result in unnecessary antibiotic use, increased length of stay, and additional laboratory tests, all of which increase healthcare costs. While the optimal skin antisepsis agent for reducing blood culture contamination is not known, the cost of various agents differs substantially.

Objective: To determine the relative rates of blood culture contamination for 3 skin antisepsis interventions - 10% povidone iodine aqueous solution (PI), 2% iodine tincture (IT) and 2% chlorhexidine gluconate in 70% isopropyl alcohol (CHG) - when used by dedicated phlebotomy teams to obtain peripheral blood cultures in adult non-ICU medical and surgical patients.

DETAILED DESCRIPTION:
A group-randomized crossover trial was conducted to test the null hypothesis of no difference in blood culture contamination rates among 3 antiseptic skin preparations. The sequence of 3 different antiseptic treatments was randomly assigned to 3 separate hospital floors, therefore in this trial cross-over occurred at the hospital floor level (not the individual patient level).

Also, it is possible for subjects to have multiple blood culture sets obtained during the study. Thus, the number of blood culture sets will not equal the number of unique subjects in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient on general medical, surgical, and cardiology floors
* Receipt of a peripheral blood draw for blood culture collection
* Blood draw performed by phlebotomy team

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3879 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laraine L. Washer, MD, Principal Investigator — University of Michigan

REFERENCES:
- [Derived] Washer LL, Chenoweth C, Kim HW, Rogers MA, Malani AN, Riddell J 4th, Kuhn L, Noeyack B Jr, Neusius H, Newton DW, Saint S, Flanders SA. Blood culture contamination: a randomized trial evaluating the comparative effectiveness of 3 skin antiseptic interventions. Infect Control Hosp Epidemiol. 2013 Jan;34(1):15-21. doi: 10.1086/668777. Epub 2012 Nov 26. PMID 23221187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please note: it is possible for a single patient to have multiple blood culture sets obtained throughout the study. Therefore, number of blood culture sets will differ from the number of unique patients.
  Also, cross-over assignment occurred at the hospital floor level - not the individual subject level.
Groups:
- CHG Then PI Then IT: 2% chlorhexidine gluconate/70% isopropyl alcohol packaged in a single 1.5 ml Frepp applicators (Enturia, Leewood KS) -- CHG
  10% povidone iodine aqueous solution packaged in a single 0.67 Sepp applicator (Enturia, Leewood KS) -- PI
  Iodine tincture (2% iodine and 2% sodium iodide diluted in 50% ethanol) packaged in a single 0.67 mL Sepp applicator (Enturia, Leewood KS) -- IT
- IT Then CHG Then PI: Iodine tincture (2% iodine and 2% sodium iodide diluted in 50% ethanol) packaged in a single 0.67 mL Sepp applicator (Enturia, Leewood KS) -- IT
  2% chlorhexidine gluconate/70% isopropyl alcohol packaged in a single 1.5 ml Frepp applicators (Enturia, Leewood KS) -- CHG
  10% povidone iodine aqueous solution packaged in a single 0.67 Sepp applicator (Enturia, Leewood KS) -- PI
- PI Then IT Then CHG: 10% povidone iodine aqueous solution packaged in a single 0.67 Sepp applicator (Enturia, Leewood KS) -- PI
  Iodine tincture (2% iodine and 2% sodium iodide diluted in 50% ethanol) packaged in a single 0.67 mL Sepp applicator (Enturia, Leewood KS) -- IT
  2% chlorhexidine gluconate/70% isopropyl alcohol packaged in a single 1.5 ml Frepp applicators (Enturia, Leewood KS) -- CHG
Period: Overall Study
Arm/Group | CHG Then PI Then IT | IT Then CHG Then PI | PI Then IT Then CHG
Started | 1421 (It is possible for the same patient to appear in multiple sequences throughout the study.) | 1410 (It is possible for the same patient to appear in multiple sequences throughout the study.) | 1379 (It is possible for the same patient to appear in multiple sequences throughout the study.)
Completed | 1421 (It is possible for the same patient to appear in multiple sequences throughout the study.) | 1410 (It is possible for the same patient to appear in multiple sequences throughout the study.) | 1379 (It is possible for the same patient to appear in multiple sequences throughout the study.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Population
Number analyzed (Participants) | 3879
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (17.9)
Sex/Gender, Customized [Number; unit: participants] — Gender data were not collected for this study
  participants
    Male | 0
    Female | 0
    Unknown | 3879

OUTCOME MEASURES:

1. Primary Outcome: Blood Culture Contamination
Description: A culture set was considered contaminated if it yielded growth of typical skin contaminants including aerobic gram positive rods, Lactobacillus sp, Propionibacterium acnes, Micrococcus sp, Bacillus sp (not B. anthracis or B. cereus), coag negative Staphylococcus, Neisseria sp (not N. meningitides or N. gonorrhoeae), or gamma-hemolytic streptococci (not Enterococcus sp) from only 1 of 2 or more blood culture sets obtained from different sites.
Time Frame: 5 days
Population: Intention to treat analyses. Please note: it is possible for a single patient to have multiple blood culture sets obtained throughout the study. Therefore, number of blood culture sets will differ from the number of unique patients.
Measure: Number; unit: blood culture sets
Units Other Than Participants: Blood culture sets
Groups:
- Chlorhexidine Gluconate (CHG_: 2% chlorhexidine gluconate/70% isopropyl alcohol packaged in a single 1.5 ml Frepp applicators (Enturia, Leewood KS) -- CHG
- Iodine Tincture (IT): Iodine tincture (2% iodine and 2% sodium iodide diluted in 50% ethanol) packaged in a single 0.67 mL Sepp applicator (Enturia, Leewood KS) -- IT
- Povidone Iodine (PI): 10% povidone iodine aqueous solution packaged in a single 0.67 Sepp applicator (Enturia, Leewood KS) -- PI
Arm/Group | Chlorhexidine Gluconate (CHG_ | Iodine Tincture (IT) | Povidone Iodine (PI)
Number analyzed (Participants) | 1429 | 1450 | 1480
Number analyzed (Blood culture sets) | 4388 | 4230 | 4286
blood culture sets | 41 | 32 | 25

ADVERSE EVENTS:
Arm/Group | CHG Then PI Then IT | IT Then CHG Then PI | PI Then IT Then CHG
Serious Adverse Events (participants affected / at risk) | 0/1421 | 0/1410 | 0/1379
Other Adverse Events (participants affected / at risk) | 0/1421 | 0/1410 | 0/1379

LIMITATIONS AND CAVEATS:
It is possible for subjects to have multiple blood culture sets obtained during the study.Thus, the # of blood culture sets will not equal the # of subjects. Also, cross-over assignment occurred at the hospital floor level - not the subject level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No